CLINICAL TRIAL: NCT06675643
Title: Digital Remote Monitoring of Immune Checkpoint Inhibitor Therapy Induced Toxicity: A Feasibility Study of the Vigilant App (Vigilant-2)
Brief Title: Digital Remote Monitoring of Immune Checkpoint Inhibitor Therapy Induced Toxicity Using the Vigilant App
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 23-011475; NCI-2024-09081 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 23-011475 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2024-11-04; First posted 2024-11-05 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Malignant Skin Neoplasm; Melanoma
MeSH Terms: conditions — Skin Neoplasms; Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational: Patients undergo standard of care treatment with ipilimumab/nivolumab and answer questions and enter symptoms in the mobile Vigilant application. Patients wearing a compatible watch have their vital signs recorded at the same time symptoms are being entered. Based on the severity of symptoms, patients may be recommended to reach out to their healthcare team or to go to the emergency room. Additionally, patients complete a survey and may have their medical charts reviewed on study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-Interventional study

SUMMARY:
This study is being done to better understand patient experiences with using a mobile application, known as Vigilant, to monitor symptoms as outpatients and to gather preliminary data on the potential clinical benefit to remote monitoring of adverse events.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Optimize the patient (Aim 1) experience of the VIGILANT app workflow. II. Gather preliminary data on the number of patients who develop Grade 3 + 4 immune-related adverse event (irAE) or require ER visit within 100 days of registration and treatment with IPI/NIVO.

OUTLINE: This is an observational study.

Patients undergo standard of care treatment with ipilimumab/nivolumab and answer questions and enter symptoms in the mobile Vigilant application. Patients wearing a compatible watch have their vital signs recorded at the same time symptoms are being entered. Based on the severity of symptoms, patients may be recommended to reach out to their healthcare team or to go to the emergency room. Additionally, patients complete a survey and may have their medical charts reviewed on study.

ELIGIBILITY:
Inclusion Criteria:

* Any skin cancer/melanoma patient starting dual [ipilimumab/nivolumab (IPI/NIVO)] immune checkpoint inhibitor (ICI) therapy

Exclusion Criteria:

* Does not meet inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with the diagnosis of skin cancer/melanoma undergoing dual ICI therapy with ipilimumab/nivolumab (IPI/Nivo) as part of regular clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-10-14 (Actual); Primary Completion 2027-03-15 (Estimated); Study Completion 2027-03-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of grade 3-4 IR-adverse events | Up to 100 days following treatment with IPI/NIVO
  Will be assessed by the number of patients who experience at least one grade 3-4 Immune-Related Adverse Events (IR-AE) within 100 days of treatment with ipilimumab/nivolumab (IPI/NIVO). Events will be self-reported using the VIGILANT app, which is being developed to help manage adverse events after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Svetomir N. Markovic, MD, PhD, Principal Investigator — Mayo Clinic; Lisa A. Kottschade, APRN, CNP, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials